CLINICAL TRIAL: NCT02532140
Title: Phase I Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of WCK 5107 Alone and in Combination With Cefepime Administered as Single IV Doses in Healthy Human Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of WCK 5107 Alone and in Combination With Cefepime
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: W-5107-101
Record Dates: First submitted 2015-08-03; First posted 2015-08-25 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
MeSH Terms: interventions — Cefepime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- WCK 5107 (Experimental): A single administration of the investigational product will be administered intravenously in 7 SAD cohorts at different dose level . The SAD cohorts will enroll 10 subjects ( 8 on active drug and 2 on placebo)
  Interventions: Drug: WCK 5107 250 mg to 2000 mg; Drug: Placebo
- WCK 5107 1000 mg and Cefepime 2000 mg (Experimental): In the crossover cohorts (WCK 5107 and cefepime, both alone and in combination), 9 subjects will receive all 3 treatments.
  Interventions: Drug: WCK 5107 250 mg to 2000 mg; Drug: Cefepime 2000 mg; Drug: WCK 5107 1000/2000 mg with Cefepime 2000 mg combination
- WCK 5107 2000 mg and Cefepime 2000 mg (Experimental): In the crossover cohorts (WCK 5107 and cefepime, both alone and in combination), 9 subjects will receive all 3 treatments.
  Interventions: Drug: WCK 5107 250 mg to 2000 mg; Drug: Cefepime 2000 mg; Drug: WCK 5107 1000/2000 mg with Cefepime 2000 mg combination

INTERVENTIONS:
Drug: WCK 5107 250 mg to 2000 mg
Drug: Cefepime 2000 mg
  Arms: WCK 5107 1000 mg and Cefepime 2000 mg; WCK 5107 2000 mg and Cefepime 2000 mg
Drug: WCK 5107 1000/2000 mg with Cefepime 2000 mg combination
  Arms: WCK 5107 1000 mg and Cefepime 2000 mg; WCK 5107 2000 mg and Cefepime 2000 mg
Drug: Placebo
  Arms: WCK 5107

SUMMARY:
• To evaluate the safety,tolerability and pharmacokinetics of single intravenous doses of WCK 5107 alone and in combination with cefepime in healthy adult human subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-55 years of age (both inclusive).
2. Have a body mass index of 18-30 kg/m2 (both inclusive) calculated as weight (kg)/height (m2).
3. Medical history without any major pathology/surgery in the last 6 months prior to screening.
4. Resting supine blood pressure of 90-139 (systolic)/40-89 (diastolic) mmHg and a resting pulse rate of 40-100 beats per minute.
5. Calculated creatinine clearance ≥80 mL/min
6. Computerized 12-lead ECG recording without signs of clinically significant pathology and showing no clinically significant deviation as judged by the Principal Investigator.
7. Males willing to use double-barrier contraceptive measures and to not donate sperm until 90 days after the follow-up visit.
8. Females should not be pregnant or breast feeding (pregnancy will be confirmed by a urine pregnancy test at screening with confirmation by a serum pregnancy test at admission) or of non-childbearing potential at screening.
9. Females must be either post-menopausal for at least 1 year, surgically sterile (bilateral oophorectomy or hysterectomy), or practicing 1 of the acceptable methods of birth control.

Exclusion Criteria:

1. History/evidence of clinically relevant pathology.
2. History of clinically significant food or drug allergy, including known hypersensitivity to cefepime or any other related drugs.
3. A positive screen result for drugs of abuse/alcohol at admission to the study center.
4. Use of prescription medications (with the exception of oral contraceptives and hormone replacement therapy) including nonsteroidal anti-inflammatory drugs or sucralfate or herbal preparations.
5. Positive screen result for hepatitis B, hepatitis C, or human immunodeficiency virus at screening.
6. Any strenuous activity within 4 days prior to admission to the study center. Strenuous being defined as any hard labor or exercise outside of a subject's usual behavior.
7. History of blood donation of more than 500 mL in the last 2 months prior to screening.
8. Current use or has used tobacco- or nicotine-containing products.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety - number of adverse events . | 14 days
  To evaluate the safety of single intravenous doses of WCK 5107 alone and in combination with cefepime in healthy adult human subjects.
Tolerability-measure of laboratory parameters | 14 days
  To evaluate the tolerability of single intravenous doses of WCK

SECONDARY OUTCOMES:
PK- Cmax | 3 days
  To evaluate the PK of single intravenous doses of WCK 5107 alone and in combination with cefepime in healthy adult human subjects.
PK-AUC | 3 days
  To evaluate the PK of single intravenous doses of WCK 5107 alone and in combination with cefepime in healthy adult human subjects.
PK-time to Cmax | 3 days
  To evaluate the PK of single intravenous doses of WCK 5107 alone and in combination with cefepime in healthy adult human subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles, Overland Park, Kansas, United States